CLINICAL TRIAL: NCT02598505
Title: Indacaterol in Heart Failure Patients: Any Role on Lung Fluid Regulation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centro Cardiologico Monzino (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Piergiuseppe Agostoni, PhD, Centro Cardiologico Monzino
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R111/14 CCM 89
Record Dates: First submitted 2015-10-22; First posted 2015-11-06 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — indacaterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Indacaterol (Experimental): Inside this arm we also compare the effect of Carvedilol to the effect of Bisoprolol
  Interventions: Drug: Indacaterol
- Placebo (Placebo Comparator): Inside this arm we also compare the effect of Carvedilol to the effect of Bisoprolol
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Indacaterol
  Arms: Indacaterol
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purposes of this study are:

1. To confirm safety of Indacaterol in stable Heart Failure.
2. To determine whether beta 2 alveolar receptor stimulation by Indacaterol is able to ameliorate lung diffusion in heart Failure patients treated with beta blockers.
3. To compare the effects of Indacaterol in patients treated with a non-selective beta blocker (Carvedilol) and a beta 1-selective beta blocker (Bisoprolol).

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults aged ≥ 18 years who have signed an Informed Consent Form.
* Patients with light chronic obstructive pulmonary disease never treated with bronchodilator drugs
* Co-operative patients
* Patients with a clinical diagnosis of chronic heart failure (HF)
* chronic myeloproliferative disorder with ejection fraction < 40% with B Blockers therapy since at least 2 months. Optimized and individually tailored drug treatment including B blocker (Carvedilol or bisoprolol)
* Capability of performing Cardiopulmonary Exercise Test and lung diffusion test

Exclusion Criteria:

History or clinical documentation of:

* pulmonary embolism
* primary valvular heart disease
* pericardial disease
* severe obstructive lung disease
* significant peripheral vascular disease
* exercise-induced angina, st changes, or severe arrhythmias.
* Patients with diabetes Type I or uncontrolled diabetes Type II including patients with a history of blood glucose levels consistently outside the normal range or HbA1c > 8.0 % of total hemoglobin measured.
* Use of bronchodilators.
* Patients with a history (or family history) of long QT syndrome or whose corrected QT interval interval (Fridericia) measured at Visit 2 is prolonged: >450 ms (males) or >470 ms (females) as assessed by the central electrocardiogram (ECG) interpretation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
measurement of change in lung diffusion of carbon monoxide (CO). | day 0, 60, 74, 134
  comparison of change in lung diffusion of carbon monoxide after treatment placebo/indacaterol between the carvedilol and bisoprolol groups.
measurement of change in membrane diffusion (Dm) | day 0, 60, 74, 134
  comparison of change in mambrane diffusion (Dm) after treatment placebo/indacaterol between the carvedilol and bisoprolol groups.
measurement of change in capillary volume (Vc) | day 0, 60, 74, 134
  comparison of change in Vc after treatment placebo/indacaterol between the carvedilol and bisoprolol groups.
measurement of change in lung diffusion of NO (Nitric Oxide) | day 0, 60, 74, 134
  Measurement of change in lung diffusion of nitric oxide after treatment placebo/indacaterol between the carvedilol and bisoprolol groups.

CONTACTS AND LOCATIONS:
Overall Officials: Piergiuseppe Agostoni, MD, Principal Investigator — Centro Cardiologico Monzino
Locations (1):
- Centro Cardiologico Monzino, Milan, MI, Italy